CLINICAL TRIAL: NCT00868998
Title: Phase II Study of the Gemzar, Taxotere and Xeloda Regimen (GTX) for Inoperable or Metastatic Adenocarcinoma of the Biliary System
Brief Title: GTX Regimen for Biliary Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor patient accrual
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB3329
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Biliary Cancer
Keywords: Biliary Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Gemcitabine, docetaxel, and capecitabine
  Interventions: Drug: Gemcitabine, docetaxel, and capecitabine

INTERVENTIONS:
Drug: Gemcitabine, docetaxel, and capecitabine — Day 1-14: Capecitabine 600 mg/m2/day (maximum dose 2000 mg/m2/day total divided into BID PO doses) Day 4 and 11: Gemcitabine 600 mg/m2 IV over 60 mins Day 4 and 11: Docetaxel 30 mg/m2 IV over 60 mins preceded by 12 mg dexamethasone IV or PO or 4 mg if diabetic
  Other Names: Gemzar; Taxotere; Xeloda

SUMMARY:
This is a study for patients with advanced cancer of the biliary tree, such as cholangiocarcinoma. They will be treated with a chemotherapy regimen consisting of Gemcitabine, Taxotere, and Xeloda every 21 days for at least 9 weeks. Treatment will continue until their cancer progresses. This chemotherapy regimen has been used in pancreatic cancer and there is reason to believe that it will be effective for cancers of the biliary tree as well.

DETAILED DESCRIPTION:
After initial presentation of our data concerning this regimen (in pancreatic cancer) at the 2003 and 2004 ASCO meetings, a number of practitioners began using the regimen for pancreatic cancer patients. More importantly, several of these investigators began using the same regimen for patients with unresectable and metastatic biliary tree cancers, such as cholangiocarcinoma. In personal communications with us, they have cited the absence of reasonable alternatives as the primary reason to experiment with novel regimens. They have described to us case reports, whereby patients with cholangiocarcinoma had objective responses to this regimen. Personally, our group, in a pilot study, has treated 5 patients with the GTX regimen, and has documented 3 partial responses and 1 stable disease in 3 patients afflicted with cholangiocarcinoma and 2 with gall bladder cancer. In this prospective study (to date 08/09), three patients have been enrolled and two of them achieved a partial response, by RECIST parameters, of >30% reduction in tumor size by cycle 3 (the first evaluation point). Therefore, we believe that GTX will show efficacy in treating this disease.

Indeed, there is clinical evidence of efficacy of these drugs in cholangiocarcinomas. In a phase II trial, single agent gemcitabine produced a 30% partial response rate and a 30% stable disease rate in chemotherapy-naïve, cholangiocarcinoma patients.(8) A retrospective review of patients treated with combination fluorouracil (continuous infusion) and gemcitabine (30 minute infusion) demonstrated a 33% response rate and a 30% stable disease rate, with a median survival of 5.3 months. The low, observed rate of grade 3-4 myelosuppression (11%) suggests this is a well tolerated regimen.(9) Likewise, gemcitabine and docetaxel have been combined in the treatment of these cancers, resulting in a 33% response rate and a 36% stable disease rate (3). We hope to improve upon these studies by substituting a sixty minute infusion rate for gemcitabine instead of the traditional thirty minute infusion, and by substituting capecitabine for infused fluorouracil. In addition, we have tested the GTX regimen in 2 cell lines in our lab: one cholangiocarcinoma and one gall bladder human line. We found that when GTX is given all at once to the cells, there is no increased cytotoxicity, but when given in the amount and dosing sequence that mimics the GTX regimen of this protocol, there is significant synergistic cytotoxicity. This synergism produces approximately a 3-fold increase in cell kill as compared with any other combination of the drugs or from any single drug in the GTX regimen. Given our laboratory data in cholangiocarcinoma cell lines that demonstrates synergy between these drugs, we are optimistic that we can produce superior results with less toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the intrahepatic or extrahepatic biliary tract including cholangiocarcinoma, gallbladder cancer and ampullary cancer (ampula of vater).
* Prior therapy with gemcitabine, Xeloda or docetaxel is acceptable if he/she only received and failed one of the 3 drugs.
* Prior experimental drug therapies such as Phase I agents are acceptable.
* Measurable disease: Any mass measurable by RECIST 1.1 parameters by CT or MRI scans of metastatic and primary tumor sites
* Ineligible for other high priority national or institutional studies
* Prior radiation and surgery allowed:

  * 3 weeks since surgery or last chemotherapy
  * 4 weeks since RT
* Non pregnant females with a negative serum β-HCG test within 1 week of starting the study, who are not breast feeding. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter.
* Clinical Parameters Life expectancy > 3 months Age ≥ 18 y.o Performance status 0-2 (ECOG) (See Appendix IV) Peripheral Neuropathy must be ≤ grade 1 Able to tolerate oral chemotherapeutic medications
* Required initial laboratory data

CBC with Differential Basic Metabolic Panel (BMP) Liver Function Tests (LFTs) Serum β-HCG (non-menopausal females) Tumor Specific Tests Hepatitis B and C Tests Pulse Oximetry on Room Air >90%

* Informed Consent: Each patient must be completely aware of the nature of his/her disease process and must willingly give consent after being informed of the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts.

Exclusion Criteria:

* Hypersensitivity: Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 must be excluded.
* Prior malignancy in last 5 years other than: curatively treated carcinoma in-situ of the cervix, non-melanoma skin cancer, DCIS (ductal carcinoma in situ) or early stage (I or II) prostate cancer previously treated with curative intent by radiation and/or surgery and is now cancer free.
* Known serious medical or psychiatric illness preventing informed consent or intensive treatment (e.g., serious infection).
* Patients with CNS metastases shall be excluded.
* Patients with compromised immune systems are at increased risk of toxicity and lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients are excluded from the study.
* Patients with currently active inflammatory bowel disease (ulcerative colitis, Crohn's) or sclerosing cholangitis will be excluded. A history of these IBD's or sclerosing cholangitis is acceptable if the disease is in remission or quiescent.
* Active infection with non-A hepatitis virus (Hepatitis B and C) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-08; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Fine, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 5
Completed | 0
Not Completed | 5
Not completed — Screen Failure | 1
Not completed — Withdrawal by Subject | 1
Not completed — Progression of disease | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants]
  50-59 | 1
  60-69 | 3
  70-79 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Data was not analyzed due to poor accrual.
Time Frame: 10 weeks
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Toxicity
Description: Data was not analyzed due to poor accrual.
Time Frame: Prior to day 4 and on day 12
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=4)
Dehydration and low blood pressure (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=4)
Bruising (General disorders) | 1 (1)
Nausea (General disorders) | 2 (2)
Vomiting (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Edema (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (General disorders) | 1 (1)
Change in taste (General disorders) | 1 (1)
Change in appetite (General disorders) | 1 (1)
Ascites (General disorders) | 1 (1)
Oral ulcer bleeding (General disorders) | 1 (1)
Mucositis (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes